# Fluid REStriction in Heart failure versus liberal fluid Uptake: the FRESH-UP study

## **Summary of changes**

| Protocol ID | NL75112.091.20 / NCT04551729 |
|---|---|
| Short title | FRESH-UP |
| First approved version | 2.0 |
| Date of first approved | 30 <sup>th</sup> November 2020 |
| version | |
| Protocol version | 3.0 |
| Date of change | 21st July 2021 |
| Section of change | Protocol information page |
| Description of change | The following was added: |
| | J.J. Herrmann MD (Radboudumc) |
| | R. Pisters MD PhD (Rijnstate) |
| Rationale for change | New coordinating investigator was added (J.J. Herrmann MD, |
| | Radboudumc, Nijmegen, The Netherlands). |
| | New including site was added (Rijnstate Hospital, Arnhem, |
| | the Netherlands). |
| Section of change | 4.3 Exclusion criteria |
| Description of change | The following criterion was added: |
| | Changes in HF medical therapy in last 14 days prior to |
| | randomization. |
| Rationale for change | To ensure within the protocol that recent pharmacological |
| | changes of the study participants could not influence baseline |
| | measurements (including Kansas City Cardiomyopathy |
| | Questionnaire (KCCQ)). |
| Section of change | 7.4 Data Safety Monitoring Board |
| Description of change | The DSMB has two mandates: |
| | 1) To perform two interim analyses at the enrolment of 33% |
| | and 66% of the subjects for safety on the occurrence of the |
| | composite clinical endpoint death, all-cause hospitalisation |
| | and the need for iv-loop diuretics; and for safety on the |
| | 1 |

occurrence of acute kidney injury; 2) To monitor the overall conduct of the trial, i.e. to monitor the enrolment rate. The above interim stage analyses will be performed for safety on two timepoints based on the number of enrolled subjects. First interim analysis will be performed at enrolment of 33% of the subjects, second at enrolment of 66% of the subjects. Was changed to: The DSMB has two mandates: 1) To perform two interim analyses when data is available at the enrolment of 33% and 66% of the subjects for safety on the occurrence of the composite clinical endpoint death, all-cause hospitalisation and the need for iv-loop diuretics; and for safety on the occurrence of acute kidney injury; 2) To monitor the overall conduct of the trial, i.e. to monitor the enrolment rate. The above interim stage analyses will be performed for safety on two timepoints based on the number of enrolled subjects. First interim analysis will be performed when data is available at the enrolment of 33% of the subjects, second when data is available at the enrolment of 66% of the subjects. To elucidate that the interim analyses will be performed when Rationale for change data from the first 33% and 66% of the study population are available. **Protocol version** 3.1 21st February 2022 Date of change Section of change Protocol information page **Description of change** The following was added: S. van Wijk MD PhD (Zuyderland Medisch Centrum)

| Rationale for change | New including site was added (Zuyderland Medisch Centrum, |
|---|---|
| | Heerlen, the Netherlands). |
| Protocol version | 4.0 |
| Date of change | 1 <sup>st</sup> June 2022 |
| Section of change | Protocol information page |
| Description of change | To be determined |
| | Was changed to: |
| | P. Van Der Meer MD PhD (chair; UMCG) |
| | Remaining members ∓to be determined |
| Rationale for change | New chair of the event adjudication committee (EAC) was |
| | added (P. Van Der Meer MD PhD (UMC Groningen, |
| | Groningen, the Netherlands). |
| Section of change | 2. Objectives |
| Description of change | Primary Objective: |
| | To investigate the effect of liberal fluid intake versus standard |
| | fluid restriction (1500cc/24hours) on QoL in outpatient |
| | chronic HF patients at 3 months after randomization, as |
| | assessed with the Kansas City Cardiomyopathy |
| | Questionnaire (KCCQ) (10) and the validated Thirst Distress Scale (11). |
| | As recently described in a "state-of-the-art-paper" in JACC: |
| | Heart Failure, the KCCQ is a well-validated questionnaire |
| | specific to HF, is sensitive to change in clinical status, and |
| | moreover, a change in KCCQ is predictive of future adverse |
| | disease progression (11, 12). |
| | For example, whereas an improvement in general well-being |
| | in terms mental health is expected to positively affect the |
| | score, any deterioration of HF is expected to negatively affect |
| | the score. Therefore, the KCCQ is perfectly suited to address |
| | both aspects of the hypothesis of this study (i.e. beneficial |
| | effects on QoL as well as signals of potential safety issues). |

In addition, the Thirst Distress Scale is most likely a sensitive measure to subtle changes in QoL due to differences in lifestyle advice concerning fluid intake.

#### Secondary Objectives:

 To investigate the effect of standard fluid restriction (1500cc/24hours) versus liberal fluid intake on QoL at 3 months after randomization, as assessed with a visual analogue scale (EQ-5D-5L);

#### Was changed to:

Primary Objective:

To investigate the effect of liberal fluid intake versus standard fluid restriction (1500cc/24hours) on QoL in outpatient chronic HF patients at 3 months after randomization, as assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ) **Overall Summary Score (OSS)** (10) and the validated Thirst Distress Scale (11).

As recently described in a "state-of-the-art-paper" in JACC: Heart Failure, the KCCQ is a well-validated questionnaire specific to HF, is sensitive to change in clinical status, and moreover, a change in KCCQ is predictive of future adverse disease progression (11, 12).

For example, whereas an improvement in general well-being in terms mental health is expected to positively affect the score, any deterioration of HF is expected to negatively affect the score. Therefore, the KCCQ is perfectly suited to address both aspects of the hypothesis of this study (i.e. beneficial effects on QoL as well as signals of potential safety issues).

In addition, the Thirst Distress Scale is most likely a sensitive measure to subtle changes in QoL due to differences in lifestyle advice concerning fluid intake.

| | Secondary Objectives: |
|---|---|
| | To investigate the effect of standard fluid |
| | restriction (1500cc/24hours) versus liberal fluid intake on |
| | thirst distress at 3 months after randomization, as |
| | assessed with TDS-HF (13); |
| | To investigate the effect of standard fluid restriction |
| | (1500cc/24hours) versus liberal fluid intake on QoL at 3 |
| | months after randomization, as assessed with by KCCQ |
| | Clinical Summary Score (CSS), each of the KCCQ |
| | domains and the proportion of patients with clinically |
| | meaningful changes in these scores and a visual |
| | analogue scale (EQ-5D-5L); |
| Section of change | 4.4 Sample size calculation |
| Description of change | The following was deleted: |
| | Both primary hypotheses on QoL by the KCCQ-OS score and |
| | thirst distress scale will be tested at a 2-sided 5% |
| | significance level. In the case of non-significant findings for |
| | the first primary end point (KCCQ), the second primary end |
| | point will be tested at the 2-sided 5% significance level but |
| | will be regarded as an exploratory end point, and a nominal P |
| | value will be produced. No adjustments for multiplicity will be |
| | made for secondary or exploratory end points. |
| Section of change | 6.1 Study parameters/endpoints |
| Description of change | 6.1.1 Main study parameters |
| | - QoL at 3 months after randomization, as assessed with the |
| | KCCQ Overall Summary (OS) Score (10) |
| | - QoL at 3 months after randomization, as assessed with the |
| | Thirst Distress Scale |
| | 6.1.2 Secondary study parameters |
| | - QoL at 3 months after randomization, as assessed with the |
| | KCCQ Clinical Summary (CS) Score and each of the KCCQ |
| | domains (10); |

| | Was changed to: |
|---|---|
| | 6.1.1 Main study parameters |
| | - QoL at 3 months after randomization, as assessed with the |
| | KCCQ Overall Summary (OSS) Score (10) |
| | -QoL at 3 months after randomization, as assessed with the |
| | Thirst Distress Scale |
| | 6.1.2 Secondary study parameters |
| | - Thirst distress at 3 months after randomization, as |
| | assessed with the TDS-HF (13) |
| | - QoL at 3 months after randomization, as assessed with the |
| | KCCQ Clinical Summary <b>Score</b> (CS <b>S</b> ) <del>Score</del> and each of the |
| | KCCQ domains (10); |
| Rationale for the three | Based on external peer and editorial review by the Journal of |
| changes above | Cardiac Failure of our "rationale-and-design-paper" and |
| | second internal statistical review, we improved the quality of |
| | our protocol accordingly. The comments and rebuttal letter |
| | are included in Appendix A. At the time of submission, and |
| | during the review process, only 140 patients were included |
| | and therefore no DSMB analysis was performed yet. |
| | Because of these changes, the primary research question |
| | how quality of life is affected by liberal fluid intake compared |
| | to fluid restriction will be answered more unambiguously. |
| | The results of the study will be easier to interpret by using |
| | one primary endpoint |
| Section of change | 4.4 Sample size calculation |
| Section of change | 4.4 Sample size calculation |
| Description of change | To test this difference at a p-value of 0.05 and power of 80%, |
| | we need a total of 454 evaluable patients. Anticipating a |
| | drop-out rate of 10% we aim to enrol 498 patients. |
| | Was changed to: |
| | To test this difference at a p-value of 0.05 and power of 80%, |
| | we need a total of 454 evaluable patients. Anticipating a |
| | drop-out rate of 10% we aim to enrol 498 <b>506</b> patients. |

| Rationale for change | To correct the inaccurate way of processing the anticipated |
|---|---|
| | 10% dropout rate in the sample size calculation using the |
| | standard LTF adjustment. |
| Section of change | 8. Statistical analysis |
| | , |
| Description of change | 8.3 Primary study parameters |
| | The difference between the two treatment arms in QoL after |
| | 3 months, as assessed with KCCQ- OS Score and Thirst |
| | Distress Score, will be tested with the use of a repeated |
| | measures ANCOVA analysis, using baseline QoL as a |
| | covariate. A p-value of <0.05 will be considered significant. |
| | Primarily, we will analyze the data for those patients, of |
| | whom both baseline and follow-up are available, similar to |
| | previous studies (16, 21). We do not expect a difference in |
| | rate of lost-to-follow-up for the primary study parameters, and |
| | rates of lost-to-follow-up will be reported for both |
| | randomization groups. |
| | We will also perform an ancillary supportive on KCCQ-OS |
| | score, in which we will give all "non-responders" at follow-up |
| | a score of 10 or 20 points below their baseline score, in case |
| | they are respectively alive or deceased. |
| | 8.4 Secondary study parameters |
| | For the secondary parameters QoL at 3 months after |
| | randomization, as assessed with the KCCQ- CS Score, each |
| | of the KCCQ domains and the EQ-5D-5L; and thirst intensity |
| | at 3 months after randomization, a similar approach as for the |
| | primary study parameters will be adopted. |
| | Was changed to: |
| | 8.3 Primary study parameters |
| | The difference between the two treatment arms in QoL after |
| | 3 months, as assessed with KCCQOS-S <del>core and Thirst</del> |
| | Distress Score, will be tested with the use of a repeated |

measures ANCOVA analysis, using baseline QoL as a covariate. A p-value of <0.05 will be considered significant.

Primarily, we will analyze the data for those patients, of whom both baseline and follow-up are available, similar to previous studiesaccording to the intention-to-treat principle (16, 21). We do not expect a difference in rate of lost-to-follow-up for the primary study parameters, and rates of lost-to-follow-up will be reported for both randomization groups.

In the unlikely case that any baseline scores on the KCCQ-OSS are missing, these will first be multiply imputed using imputations drawn from the distribution of the full study population. Following this, the imputation model will be specified separately by treatment arm and will include baseline and 3-month KCCQ-OSS as well as any auxiliary variables that are considered to be associated with the outcome or with the probability of missing the 3-month KCCQ scores.

We will also perform an ancillary sensitivity supportive analysis to examine the sensitivity of the results to missing data assumptions on KCCQ-OS score, in which we will give all "non-responders" at follow-up a score of 10 or 20 points below their baseline score, in case they are respectively alive or deceased. For this sensitivity analysis, a delta-adjustment approach will be applied, with a fixed constant (to be elicited from a panel of experts) added to the values imputed under the standard MAR procedure (22).

### 8.4 Secondary study parameters

For the secondary parameters **thirst distress**, **as assessed** with the TDS-HF, and QoL at 3 months after randomization, as assessed with the KCCQ--CS-Score, each of the KCCQ domains and the EQ-5D-5L; and thirst intensity at 3 months

| | after randomization, a similar approach as for the primary |
|---|---|
| | study parameters will be adopted. |
| | Stady parameters will be adopted. |
| Rationale for change | To emphasize that the intention-to-treat method will be used |
| | for the primary analysis as described in paragraph 8.2. |
| | To increase the generalizability of the possible imputed |
| | missing baseline scores, the single imputation method was |
| | changed to a multiple imputation method. However, since |
| | quality of life measurements are known to be missing not at |
| | random, a sensitivity analysis was included. |
| Section of change | DSMB Charter; Annex 3: interim analysis |
| Description of change | The following will be the main parameters of interest for the |
| | DSMB: |
| | KCCQ scores |
| | The occurrence of HF hospitalizations |
| | The occurrence of death |
| | The occurrence of acute kidney injury |
| | These data will be made available to the DSMB before to the |
| | interim analyses, should be explicitly discussed and reported |
| | by the DSMB in their reports. |
| | 2, and 20m2 in alon reporter |
| | This trial aims to include 498 patients. The first interim |
| | analysis by the DSMB will be performed when data is |
| | available on 33% of patients and the second when data is |
| | available on 66% of patients. Possible recommendations |
| | after the interim analysis could include, but are not exclusive |
| | to: |
| | No action needed, trial continues as planned |
| | · |
| | Early stopping due to harm of a treatment or clear auppriority |
| | superiority Senetianing and/or proposing protocol changes such |
| | Sanctioning and/or proposing protocol changes, such |
| | as a change in sample size in case of large discrepancies |
| | between expected and observed event rates in the control |
| | arm. |
| | Was changed to: |

| | The following will be the main parameters of interest for the |
|---|---|
| | DSMB: |
| | <ul> <li>KCCQ scores</li> <li>The occurrence of HF hospitalizations</li> <li>The occurrence of death</li> <li>The occurrence of acute kidney injury</li> </ul> |
| | These data will be made available to the DSMB before to the interim analyses, should be explicitly discussed and reported by the DSMB in their reports. |
| | This trial aims to include 498506 patients. The first interim analysis by the DSMB will be performed when data is available on 33% of patients and the second when data is available on 66% of patients. Possible recommendations after the interim analysis could include, but are not exclusive to: No action needed, trial continues as planned Early stopping due to harm of a treatment or clear superiority Sanctioning and/or proposing protocol changes, such as a change in sample size in case of large discrepancies between expected and observed event rates in the control arm. |
| Rationale for change | To clarify that the DSMB only can make recommendations to the investigators concerning continuation, termination, or other modifications of the study based on safety and not efficacy. |
| Protocol version | 4.1 |
| Date of change | 29 <sup>th</sup> September 2022 |
| Section of change | Protocol information page |
| Description of change | The following was added: J.W.M. Van Eck MD PhD MSc (Jeroen Bosch Ziekenhuis) |

| Rationale for change | New including site was added (Jeroen Bosch Hospital, Den |
|---|---|
| | Bosch, the Netherlands). |
| Section of change | Protocol information page |
| Description of change | The following was added: |
| | F.H. Verbrugge MD PhD (UZ Brussel, België) |
| | M.L. Handoko MD PhD (Amsterdam UMC) |
| Rationale for change | New members of the EAC were added (F.H. Verbrugge MD |
| | PhD (UZ Brussel, Belgium) and M.L. Handoko MD PhD |
| | (Amsterdam UMC, Amsterdam, The Netherlands)). |
| Protocol version | 4.2 |
| Date of change | 2 <sup>nd</sup> December 2022 |
| Section of change | Protocol information page |
| Description of change | The following was added: |
| | G.C.M. Linssen MD PhD (Ziekenhuisgroep Twente) |
| Rationale for change | New including site was added (Ziekenhuisgroep Twente, |
| | Almelo, the Netherlands). |
| Protocol version | 4.3 |
| Date of change | 5 <sup>th</sup> December 2023 |
| Section of change | Protocol information page |
| Description of change | The following was added: |
| | S.C.A.M. Bekkers MD PhD (Bernhoven Ziekenhuis) |
| Rationale for change | New including site was added (Bernhoven Hospital, Uden, |
| | the Netherlands). |
| Protocol version | 4.4 |
| Date of change | 15 <sup>th</sup> May 2024 |
| Section of change | Protocol information page |
| Description of change | The following was added: |
| | E. Wierda MD LLM PhD (Dijklander Ziekenhuis) |

| Rationale for change | New including site was added (Dijklander Hospital, Hoorn, |
|---|---|
| | the Netherlands). |